CLINICAL TRIAL: NCT07331051
Title: The Relationship Between Nutritional Attitudes and Anthropometric Measurements and Agility in Elite Football Players
Brief Title: Nutritional Attitudes and Anthropometric Measurements in Relation to Agility in Football Players
Status: Completed | Type: Observational
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Neslihan Altuntas Yilmaz, Principal Investigator, Necmettin Erbakan University
Other Study IDs: NEU-PT2025-03
Record Dates: First submitted 2025-12-15; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Healthy Adolescent Soccer Players
Keywords: Agility; Body composition; Anthropometric measurements; Nutritional attitudes; Adolescent soccer players; Football performance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy adolescent soccer players: This cohort consists of healthy adolescent soccer players aged 14-18 years who have been playing at club level for at least three years and have regularly participated in a minimum of four training sessions per week. This is an observational, cross-sectional study with no intervention applied. Sociodemographic characteristics, nutritional attitudes, anthropometric measurements, body composition, and agility performance were assessed.

SUMMARY:
Soccer players' agility can be affected by many factors, including nutrition and body composition. The primary objective of our study is to reveal the relationship between nutritional attitudes and anthropometric measurements and agility in elite adolescent soccer players. Our secondary objective is to determine the effect of daily fluid intake and daily sleep duration on anthropometric measurements, nutrition attitude scores, and agility in soccer players. Study was conducted on 51 male soccer players aged 14-18. Information on the soccer players' sociodemographic characteristics and lifestyles was obtained via a questionnaire. Body composition analysis was measured using a Bioelectrical Impedance Analysis (BIA) device, and hand grip strength was measured using a hand grip dynamometer. Height, waist circumference, and hip circumference were measured. Soccer players' attitudes toward nutrition were assessed using the Nutrition Attitude Scale (NAS), and their agility was assessed using the Agility T-Test.

DETAILED DESCRIPTION:
This descriptive cross-sectional study was conducted between January 15 and March 1, 2024, with adolescent football players from the Tümosan Konyaspor Football Club. Sample size calculation was performed using G*Power 3.1.9.4 based on a correlation coefficient of 0.35, 95% power, and a 0.05 alpha level, resulting in a minimum required sample size of 41 participants. A total of 51 male football players aged 14-18 years were included.

Data were collected through face-to-face interviews using a structured questionnaire comprising sociodemographic and lifestyle characteristics, anthropometric measurements, agility assessment, and the Nutrition Attitude Scale (NAS). Anthropometric measurements and body composition parameters were assessed using bioelectrical impedance analysis, while height, waist and hip circumferences, and hand grip strength were measured using standardized procedures. Nutritional attitudes were evaluated with the NAS. Agility performance was assessed using the Agility T-test with electronic timing.

Statistical analyses were performed using SPSS version 22.0. Descriptive statistics were calculated, normality was assessed, and appropriate parametric and non-parametric tests were applied. Relationships between variables were examined using Pearson correlation analysis, with statistical significance set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 14-18 years
* At least 3 years of club-level football experience
* Regular participation in a minimum of 4 training sessions per week (excluding matches) over the past year
* Voluntary participation with written informed consent obtained from the participant and/or legal guardian

Exclusion Criteria:

* Presence of any systemic disease affecting nutritional status
* Locomotor pain or musculoskeletal conditions preventing evaluation
* Failure to obtain participant and/or parental consent

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Only male adolescent soccer players were eligible to participate in this study.
Study Population: The study population consists of healthy male adolescent soccer players aged 14-18 years who have been playing at club level for at least three years and regularly participate in a minimum of four training sessions per week.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-03-15 (Actual)

PRIMARY OUTCOMES:
Sociodemographic and lifestyle information | Baseline (single assessment).
  Sociodemographic and lifestyle information, including age, education level, disease status, smoking and alcohol use, fluid consumption, and sleep duration, will be collected using a structured questionnaire and reported descriptively as a single composite dataset.Unit of Measure:
  Composite descriptive variables
Hand grip strength | Baseline (single assessment).
  Hand grip strength was measured using a TAKEI T.K.K 5401 (Japan) brand hand grip dynamometer. During the measurement, the football players were asked to sit down with their elbows bent to the side at a 90° angle and squeeze the tool with all the hand strength they could (Massy-Westropp et al., 2011). Each hand grip strength trial lasted at least 4 seconds, with a 20-second rest period between trials (Valenzuela et al., 2020). Hand grip strength measurement was repeated twice on the right and left hands, and the highest measurements for each hand were determined and averaged to calculate hand grip strength.
Agility assessment | Baseline (single assessment).
  The agility assessment was performed by the researcher physiotherapist. The agility T-test is a running test in which four cones are arranged in a T-shape. Three cones were placed 4.57 m apart in a straight line, with the starting cone 9.14 m away, lying perpendicular to the middle cone. Football players were asked to accelerate to touch the base of each cone and to run forward, laterally, and backward between the cones as fast as possible. An electronic timer was used to record times in the test

SECONDARY OUTCOMES:
Body Fat Mass | Baseline (single assessment).
  Body fat mass was measured using a TANITA BC-418 MA (Tokyo, Japan) Bioelectrical Impedance Analysis (BIA) device with a sensitivity of 0.1 kg.
Body Weight | Baseline (single assessment)
  Body weight was measured using a calibrated scale.
Nutritional attitudes | Baseline (single assessment)
  Nutrition Attitude Scale. This scale, applied to high school and university students aged 12-25, assesses individuals' attitudes toward nutrition in relation to their consumption of processed foods, carbohydrates, vitamins, minerals, protein, and water
Body Muscle Mass | Baseline (single assessment)
  Body muscle mass was measured using a TANITA BC-418 MA (Tokyo, Japan) Bioelectrical Impedance Analysis (BIA) device with a sensitivity of 0.1 kg.
Body Water Mass | Baseline (single assessment)
  Body water mass was measured using a TANITA BC-418 MA (Tokyo, Japan) Bioelectrical Impedance Analysis (BIA) device with a sensitivity of 0.1 kg.
Body Mass Index (BMI) | Baseline (single assessment)
  Body mass index was calculated by dividing body weight (kg) by the square of height (m²).
Waist Circumference | Baseline (single assessment)
  Waist circumference was measured using a non-elastic measuring tape.
Hip Circumference | Baseline (single assessment)
  Hip circumference was measured using a non-elastic measuring tape.Unit of Measure: cm

CONTACTS AND LOCATIONS:
Overall Officials: neslihan altuntaş yılmaz, Assistant Professor, Study Director — Necmettin Erbakan University
Locations (1):
- Tumosan sports club, Konya, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared to protect participant confidentiality and privacy, as co